CLINICAL TRIAL: NCT05738837
Title: A Phase III Randomized Wait-list Controlled Trial of the Efficacy of the Adolescent Adaptation of the EAAA Sexual Assault Resistance Education Program
Brief Title: An Evaluation of a Sexual Assault Resistance Program for Adolescent Girls
Acronym: SARE-A
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Windsor (Other)
Collaborators: Public Health Agency of Canada (PHAC) (Other Government)
Responsible Party: Principal Investigator, Dr. Charlene Y. Senn, Distinguished University Professor, University of Windsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1819-HQ-000057
Record Dates: First submitted 2023-02-12; First posted 2023-02-22 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Sexual Assault
Keywords: intervention; adolescents; sexual assault; rape; dating violence; gender-based violence; girls' health; prevention

STUDY DESIGN:
Intervention Model Description: Approximately 900 self-identified girls/young women age 14-18 (who have not already graduated high school) will be recruited from 3 communities in Ontario over two years. Participants will be randomly assigned to either receive the A-EAAA program immediately (treatment group) or 6 months later (waitlist control group). Control group participants will attend a brief 'usual care' session providing them with basic information on SV and consent in parallel with the treatment group's first session. All participants will complete surveys at 4 timepoints: baseline, 1-week post-intervention (control group matched to treatment group timing), and 6 and 12 months after baseline. The control group will take the A-EAAA program following the 6-month post-survey and complete one additional survey, 1-week after their final program session.
Masking Description: All participants are blind to allocation at baseline assessment. Randomization occurs after in-person survey completion and is initially masked (using colour coded room assignments). Allocation is revealed to participants by intervention staff once they arrive at their assigned intervention room. All data analysis is done by a Co-I who has no contact with participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A-EAAA (Adolescent Enhanced Assess, Acknowledge, Act) immediately (Experimental): Adolescent adaptation of EAAA sexual assault resistance education (4, 3-hr sessions) begun immediately after baseline randomization
  Interventions: Behavioral: A-EAAA Sexual Assault Resistance Education Program immediately
- Waitlist Control (Active Comparator): Usual care 30-min session (brief presentation on consent/sexual assault; access to local resource pamphlets) immediately after baseline randomization; A-EAAA (4, 3-hr sessions) at 6-months post-randomization
  Interventions: Behavioral: Usual care + A-EAAA at 6 months

INTERVENTIONS:
Behavioral: A-EAAA Sexual Assault Resistance Education Program immediately — Adapted from the EAAA program created for university women, A-EAAA is designed for teen girls of all sexual identities and experience levels. It focuses on resisting sexual assault (SA) committed by male acquaintances with 4, 3-hour units: Unit 1(Assess) strengthens girls' ability to detect risk in contexts involving male acquaintances and helps develop strategies to reduce it. Unit 2(Acknowledge) helps girls explore ways to overcome their own emotional barriers preventing them from acknowledging risk and employing effective resistance strategies with males they know. Unit 3(Act) provides evidence on effectiveness of various resistance strategies and teaches verbal and physical self-defense focused on common acquaintance SA situations. Unit 4 (Relationships&Sexuality) is an adaptation of Our Whole Lives curriculum and aims to increase girls' comfort talking about sex/sexuality and identify their sexual values/desires and explore possibilities for sexual practices beyond intercourse.
  Other Names: Girls -- Flip the Script with EAAA
  Arms: A-EAAA (Adolescent Enhanced Assess, Acknowledge, Act) immediately
Behavioral: Usual care + A-EAAA at 6 months — Participants assigned to the waitlist control group will immediately receive a brief educational session on sexual assault that represents the current 'standard of care' at Canadian high schools (often presented by local Sexual Assault Centres or Public Health nurses). This 30-min session will involve a brief 15 - 20-minute presentation on sexual consent, respect in relationships, and sexual assault (e.g., definitions, prevalence statistics). This will be conducted by a well-trained and knowledgeable Research Assistant. Following the presentation, participants will be invited to take and read brochures provided on sexual assault, and to ask questions about the content of the presentation and brochures. At 6-months, participants will be scheduled to receive A-EAAA.
  Arms: Waitlist Control

SUMMARY:
Sexual violence (SV) perpetrated by dating partners and male acquaintances is common among adolescent girls in high school. Girls and young women who experience SV are likely to encounter negative mental and physical health consequences as well as lowered academic performance. While educational interventions to address the problem of SV are numerous, when evaluated, few show any capacity to reduce sexual violence victimization or perpetration. The Enhanced Assess, Acknowledge, Act (EAAA) sexual assault resistance program for female university students (ages 17-24) is a rare exception; in a rigorous trial, EAAA reduced attempted and completed rape by 50% in the following year. The current randomized controlled trial (RCT) will test whether a version of EAAA that has been adapted for younger girls (age 14-18) who have not graduated high school (called the Adolescent Enhanced Assess, Acknowledge, Act [A-EAAA]) will result in similar benefits within a 6-month follow-up. The current RCT will be conducted across three sites in Ontario, Canada.

DETAILED DESCRIPTION:
Sexual violence (SV), which occurs along a continuum from unwanted sexual contact to rape, is common among adolescent girls and young women: research suggests 1 in 7 teen girls experiences SV. Perpetrators of SV are overwhelmingly male; however, the programs that exist to address boys'/men's perpetration are not sufficiently effective nor are they widely available. Other approaches to sexual assault prevention for adolescents, such as bystander programs, have not been shown to reduce sexual violence victimization or perpetration. Given the numerous negative consequences associated with SV, developing effective SV prevention and resistance programs targeting teens is critical for reducing victimization and improving health outcomes for adolescent girls. The Enhanced Assess, Acknowledge, Act (EAAA) sexual assault resistance program has been shown to substantially reduce rates of SV (50% for rape and attempted rape) in young women attending university (ages 17-24), but since it was designed for university students in a different developmental stage, an evidence-based adaptation was necessary. The purpose of the current study is to test the efficacy of the newly adapted Adolescent Enhanced Assess, Acknowledge, Act (A-EAAA) program in reducing sexual violence victimization among adolescent girls within 6-months of trial entry. We will continue to follow participants for one-year to evaluate whether changes in tertiary outcomes (e.g., mediators) are maintained to 12-months. A-EAAA is a 12-hour psychoeducational intervention that provides information, skills, and practice aimed at a) decreasing the time needed for girls to assess sexually coercive situations as dangerous and to take action, b) reducing emotional obstacles to taking action, c) increasing the use of the most effective methods of verbal and physical self-defense, and d) identifying sexual and relationship values and boundaries and reinforcing the right to defend them.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified girls aged 14 to 18 years;
* have not graduated high school;
* competence in spoken and written English;
* provide informed consent;
* able to attend one of the scheduled programs in the data collection period in which they are enrolled.

Exclusion Criteria:

None

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — individuals must self-identify as girls/young women
Enrollment: 900 (Estimated)
Dates: Start 2023-03-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Completed Rape | Six months after randomization
  The Sexual Experiences Survey Short Form Victimization (SES-SFV) will be used to measure the primary sexual assault outcomes. Completed rape will have occurred when a participant indicates she has had at least one experience of threatened, forced, or drugged completed (not attempted) sexual activity (oral, anal, or vaginal intercourse - answered 'once' or more to any of 9 questions (2c, 2d, 2e, 3c, 3d, 3e, 4c, 4d, or 4e) in the period between the baseline measurement and the 6-month survey measurement.

SECONDARY OUTCOMES:
Attempted Rape | Six months after randomization
  The SES-SFV will also be used to measure secondary sexual assault outcomes: Attempted rape will have occurred when a participant indicates she has had at least one experience of threatened, forced, or drugged attempted (not completed) sexual activity (oral, anal, or vaginal intercourse - answered 'once' or more to any of 9 questions (5c, 5d, 5e, 6c, 6d, 6e, 7c, 7d, or 7e) in the period between the baseline and the 6-month survey.

OTHER OUTCOMES:
Other Forms of Sexual Assault | Six months after randomization
  The SES-SFV will also be used to measure tertiary sexual assault outcomes:
  1. Non-penetrative forced sexual contact will have occurred when a participant indicates she has had at least one such experience of non-penetrative sexual contact by any perpetrator strategy - answered 'once' or more to any of 5 questions (1a, 1b, 1c, 1d, 1e).
  2. Completed sexual coercion will have occurred when a participant indicates she has had at least one experience of coerced (not forced) completed sexual activity (oral, anal, or vaginal intercourse - answered 'once' or more to any of 6 questions (2a, 2b, 3a, 3b, 4a, 4b).
  3. Attempted sexual coercion will have occurred when a participant indicates she has had at least one experience of coerced (not forced) attempted (not completed) sexual activity (oral, anal, or vaginal intercourse - answered 'once' or more to any of 6 questions (5a, 5b, 6a, 6b, 7a, 7b).
Self-Defense Self-Efficacy | 1-week post-intervention, six months after randomization
  Measured with a questionnaire adapted by Senn et al. (2011) from Marx, Calhoun, Wilson, & Meyerson (2001) will be used to assess changes from baseline in girls' confidence that they could defend themselves if confronted with a sexual assault situation.
Perception of Personal Risk | 1-week post-intervention, six months after randomization
  A single item adapted from Gray, Lesser, & Brounds (1990) will be used to measure girls' and young women's perception of their personal risk of sexual assault by male acquaintances.
Detection of Risk Cues | 1-week post intervention, 6-months
  Scenario measures will be used to assess participants' ability to detect risk in hypothetical acquaintance scenarios. At 1-week post-intervention (measure adapted from Testa et al. (2006)), at 6- -months (acquaintance scenario adapted from Messman-Moore & Brown (2006)). Each measure can only be used once.
Knowledge/Willingness to use Effective Self-Defense Strategies | 1-week post-intervention, six months after randomization
  Direct Resistance subscale of Testa et al. (2006)'s measure used at 1-week post intervention. A survey adapted from Senn, Gee, & Thake (2011) will be used to measure changes from baseline in participants' knowledge of the most effective self-defense strategies.
Rape Beliefs | 1-week post-intervention, six months after randomization
  The Updated Illinois Rape Myth Acceptance scale (Payne et al., 1999; McMahon & Farmer, 2011), the Perceived Causes of Rape scale (Cowan & Campbell, 1995; Cowan & Quinton, 1997), and the Attitudes Toward Male Sexual Violence scale (Prince et al., 1999) will be used to measure girls' beliefs about rape.
Experience of Embodiment | 1-week post-intervention, six months after randomization
  Girls' sense of embodiment (i.e., the extent to which they feel in tune and comfortable with their bodies), measured via Piran & Teall (2012)'s questionnaire.
Self-Blame Following Sexual Assault | six months after randomization
  Behavioral self-blame subscale from Frazier et al. (2005) will be used to assess the extent to which girls who are sexually assaulted in the follow-up timeframe of the trial blame themselves for the incident(s).

CONTACTS AND LOCATIONS:
Overall Officials: Charlene Y Senn, PhD, Principal Investigator — University of Windsor; Sara E Crann, PhD, Principal Investigator — University of Windsor
Locations (1):
- University of Windsor, Windsor, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers will be allowed to access de-identified survey responses upon request to the PIs.
Supporting Information: Study Protocol, SAP
Time Frame: from first publication (estimated 2026) for 5 years.
Access Criteria: Request submitted to one of the PIs from qualified university researcher.

REFERENCES:
- [Background] Senn CY, Eliasziw M, Barata PC, Thurston WE, Newby-Clark IR, Radtke HL, Hobden KL. Efficacy of a sexual assault resistance program for university women. N Engl J Med. 2015 Jun 11;372(24):2326-35. doi: 10.1056/NEJMsa1411131. PMID 26061837
- [Background] Senn CY, Eliasziw M, Hobden KL, Newby-Clark IR, Barata PC, Radtke HL, Thurston WE. Secondary and 2-Year Outcomes of a Sexual Assault Resistance Program for University Women. Psychol Women Q. 2017 Jun;41(2):147-162. doi: 10.1177/0361684317690119. Epub 2017 Mar 2. PMID 29503496